CLINICAL TRIAL: NCT03655743
Title: Development of a New Patient Reported Outcome (PRO) Measure for Refractive Surgery Patients as Part of the National Dataset in Refractive Surgery
Brief Title: PRO Measure for Refractive Surgery IRAS Project Number 246072
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ALLB1020
Record Dates: First submitted 2018-08-10; First posted 2018-08-31 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Refractive Errors; Satisfaction; Cornea; Lens Diseases
MeSH Terms: conditions — Refractive Errors; Personal Satisfaction; Corneal Diseases; Lens Diseases | interventions — Keratomileusis, Laser In Situ; Photorefractive Keratectomy; Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients after refractive surgery: Patients have had any type of corneal or lens refractive surgery.
  Interventions: Device: LASIK, PRK, Phacoemulsification
- Patients before refractive surgery: Patients will have any type of corneal or lens refractive surgery.
  Interventions: Device: LASIK, PRK, Phacoemulsification

INTERVENTIONS:
Device: LASIK, PRK, Phacoemulsification — Please see:
  https://en.wikipedia.org/wiki/LASIK https://en.wikipedia.org/wiki/Photorefractive_keratectomy https://en.wikipedia.org/wiki/Phacoemulsification

SUMMARY:
The development and validation of a concise, practical, on-line, self-administered, self-archiving, and self-scoring PRO questionnaire for routine clinical use in refractive surgery is the primary study objective. Secondary objectives are to gather outcome data from patients before and after surgery in each of the following domains comprising key elements of vision related quality of life: spectacle dependence; quality of vision; eye comfort; freedom; emotional well-being; and overall satisfaction with the results of surgery. Patients undergoing refractive surgery at Moorfields Private Outpatient Clinic will be enrolled in the study in the validation phase.

DETAILED DESCRIPTION:
Specific aims of the study The investigators aim to take a novel PRO questionnaire from the conceptual framing stage through a well-defined validation pathway including cognitive interviews, field data collection in the target population, and Rasch modification. Secondary aims are to take the modified instrument through prospective studies of repeatability and sensitivity to change. The investigators´ ultimate goal is to develop a concise, screen based, self-administered, self-archiving and self-scoring PRO instrument for use as part of the National Dataset in Refractive Surgery.

Study Design

Step 1. Conceptual framing and draft development Conceptual framing and draft development for the questionnaire is complete. This was based on a comprehensive literature review, patient and surgeon feedback during RCOphth Refractive Surgery Standards development consultation, and advice from a panel of expert collaborators.

The investigators began with a literature review of existing refractive error specific questionnaires, including the following: (1) National Eye Institute Refractive Quality of Life (NEI-RQL), (2) Refractive Status and Vision Profile (RSVP), (3) Quality of Life Impact of Refractive Correction (QIRC), (4) Quality of Vision (QoV), (5) Canadian Refractive Surgery Research Group Quality of Vision Questionnaire (QVQ), (6) PERK Study Questionnaire, (7) Multidimensional Quality of Life for Myopia (MQLM) Scale, (8) Myopia-Specific Quality of Life Questionnaire (MQLQ), (9) Subjective Vision Questionnaire (SVQ), (10) Refractive Error Quality of Life Scale (REQ-Thai), (11) The Freedom from Glasses Value Scale (FGVS), (12) Near Activity Visual Questionnaire (NAVQ), Catquest questionnaire (CatQuest 9SF), and ocular comfort index (OCI).

Those questionnaires have been identified as refractive error specific in a recent review article published in JRS. The ocular comfort index (OCI) addresses ocular surface irritation. Unlike previous instruments designed to measure eye comfort such as the widely used ocular surface disease index (OSDI), it is unidimensional and was developed using Rasch fitting.

According to FDA recommendations, a conceptual framework is helpful in guiding the development of a PRO instrument . Following these recommendations, the investigators first identified the aspects of PRO for refractive surgery to be measured. Each of these aspects or "domains" is measured by a set of items. The investigators identified and included the following subscales:

* Spectacle dependence
* Quality of vision
* Ocular comfort symptoms /Eye comfort (Eye comfort is used in the questionnaire)
* Freedom
* Looking and Feeling Well
* Overall satisfaction

Having defined the domains of interest, the next task was to reduce and adapt the pool of candidate questionnaire items. Winnowing refers to reducing the item pool to the smallest number of items, making sure that the domain of interest will still be adequately measured. DeWalt et al. stated that winnowing helps to accurately define and identify those item characteristics relevant to each domain. Items are deleted if they are considered to duplicate the information captured, or if they are deemed to be potentially confusing to respondents. The investigators focused preferentially on items from Rasch weighted instruments. The investigators also reviewed items within each domain attempting to ensure, with input from patients and experts, that the most relevant aspects of each domain are captured by the item sets in the draft instrument. The investigators intended to keep a set of non-redundant items that are consistent with the domain, universally understood, and relevant to a wide range of the adult population. Items were revised so they would be understood by the largest possible number of people. In addition, consistency was sought to the extent possible in wording, recall interval, and response options.

The investigators opted to use four response options based on a balance between parsimony and adequate sampling. Both the most widely used current instruments (QIRC and CatQuest), after Rasch modification in development, focus on four response option scales.

To make items more universally understood, slight modifications to item stems and/or response options from their original form were made in those cases where we believed simplification was necessary. All changes in wording were then tested versus original versions in cognitive interviews. Items that were too long or confusing were shortened.

Step 2. Cognitive interviews Cognitive interviews will be conducted to optimise face validity (comprehensibility) of items and response options. Forty participants will be recruited from the waiting rooms of the Refractive Surgery Service at Moorfields Private Eye Hospital (Consultant Bruce Allan MD). The sample should include 20 males and 20 females of different age and educational background (highest degree). A trained interviewer (Andreas Frings MD) will conduct all of the cognitive interviews. Participants will be asked to describe in their own words what each item is asking, and in some cases to compare different ways of asking the same question. These interviews will be helpful because subjects can directly provide input and suggestions on every item considered for inclusion. As a result of these interviews, items could be further simplified, some words could be deleted, some items could be reworded, and some parts of the stems could be added to response options for clarity. The revised survey will then be used for field testing.

Step 3. Field testing and item calibration After questionnaire refinement resulting from cognitive interviews, the investigators will gather completed questionnaire data from a representative cross-section of the target patient population for Rasch fitting. Step 2 is the major component of the validation study and is described in detail below.

ELIGIBILITY:
Inclusion Criteria:

Refractive Surgery

Exclusion Criteria:

Participation denied.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are planning are have had refractive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Subjective satisfaction with treatment and treatment results. | 12 months
  1. Spectacle dependence:
     Grading:
     NEVER OCCASIONALLY SOME OF THE TIME MOST OF THE TIME
  2. Quality of vision :
     Grading:
     NO PROBLEM MILD MODERATE SEVERE
  3. Ocular comfort symptoms /Eye comfort:
     Grading:
     NO PROBLEM MILD MODERATE SEVERE
  4. Freedom:
     Grading:
     NO PROBLEM MILD MODERATE SEVERE
  5. Looking and Feeling Well:
     Grading but no definitions:
     NEVER OCCASIONALLY SOME OF THE TIME MOST OF THE TIME
  6. Overall satisfaction:
  Grading:
  VERY DISSATISFIED DISSATISFIED SATISFIED VERY SATISFIED

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry S, Mangione CM, Lindblad AS, McDonnell PJ. Development of the National Eye Institute refractive error correction quality of life questionnaire: focus groups. Ophthalmology. 2003;110:2285-2291 // Bland JM & Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res 1999; 8: 135-160 // Bottomley A, Jones D, Claassens L. Patient-reported outcomes: assessment and current perspectives of the guidelines of the Food and Drug Administration and the reflection paper of the European Medicines Agency. Eur J Cancer. 2009;45:347-53 // Bourque LB, Cosand BB, Drews C, Waring GO 3rd, Lynn M, Cartwright C. Reported satisfaction, fluctuation of vision, and glare among patients one year after surgery in the Prospective Evaluation of Radial Keratotomy (PERK) Study. Arch Ophthalmol. 1986;104:356-363 // Brunette I, Gresset J, Boivin J-F, Boisjoly H, Makni H. Function¬al outcome and satisfaction after photorefractive keratectomy: Part 1. Development and validation of a survey questionnaire. Ophthalmology. 2000;107:1783-1789 // Buckhurst PJ, Wolffsohn JS, Gupta N, Naroo SA, Davies LN, Shah S. Development of a questionnaire to assess the relative subjective benefits of presbyopia correction. J Cataract Refract Surg. 2012;38:74-79 // DeWalt DA, Rothrock N, Yount S, Stone AA; PROMIS Cooperative Group. Evaluation of item candidates: the PROMIS qualitative item review. Med Care. 2007;45:12-21 // Erickson DB, Stapleton F, Erickson P, du Toit R, Giannako¬poulos E, Holden B. Development and validation of a multi¬dimensional quality-of-life scale for myopia. Optom Vis Sci. 2004;81:70-81 // Finger RP, Fenwick E, Owsley C, Holz FG, Lamoureux EL. Visual functioning and quality of life under low luminance: evaluation of the German Low Luminance Questionnaire. Invest Ophthalmol Vis Sci. 2011;52:8241-9 // Fraenkel G, Comaish lF, Lawless MA, Kelly MR, Dunn SM, Byth K, Webber SK, Sutton GL, Rogers CM. Development of a questionnaire to assess subjective vision score in myopes seeking refractive surgery. J Refract Surg. 2004;20:10-9 // Gothwal VK, Reddy SP, Bharani S, Bagga DK, Sumalini R, Garudadri CS, Rao HL, Senthil S, Pathak-Ray V, Mandal AK. Impact of glaucoma on visual functioning in Indians. Invest Ophthalmol Vis Sci. 2012;53:6081-92 // Hays RD, Mangione CM, Ellwein L, Lindblad AS, Spritzer KL, McDonnell PJ. Psychometric properties of the National Eye Institute-Refractive Error Quality of Life instrument. Ophthalmology. 2003;110:2292-301 // Johnson ME, Murphy PJ. Measurement of ocular surface irritation on a linear interval scale with the ocular comfort index (OCI). Invest Ophth Vis Sci 2007;48:4451-8 // Kandel H, Khadka J, Lundström M, Goggin M, Pesudovs K. Questionnaires for Measuring Refractive Surgery Outcomes. J Refract Surg. 2017;33:416-424 // Khadka J, McAlinden C, Pesudovs K. Quality assessment of ophthalmic questionnaires: review and recommendations. Optometry and Vision Science 2013; 90: 720-744 // Lee J, Lee J, Park K, Cho W, Kim JY, Kang HY. Assessing the value of laser in situ keratomileusis by patient-reported outcomes using quality of life assessment. J Refract Surg. 2005;21:59-71 // Lévy P, Elies D, Dithmer O, Gil-Campos I, Benmedjahed K, Berdeaux, Arnould B. Development of a new subjective questionnaire: the Freedom from Glasses Value Scale (FGVS). J Refract Surg. 2010;26:438-46 // Lundström M, Pesudovs K. Catquest-9SF: patient outcomes questionnaire - nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cat Refract Surg 2009;35:504-13 //
- [Background] Lundström M, Pesudovs K. Questionnaires for measuring cataract surgery outcomes. J Cataract Refract Surg. 2011;37:945-59 // McAlinden C, Pesudovs K, Moore JE. The development of an in¬strument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010;51:5537-5545 // Mokkink LB, Terwee CB, Knol DL, Stratford PW, Alonso J, Patrick DL, Bouter LM, de Vet HC. The COSMIN checklist for evaluating the methodological quality of studies on measurement properties: a clarification of its content. BMC Med Res Methodol 2010;10:22 // Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010;19:539-49 // Mullin PA, Lohr KN, Bresnahan BW, McNulty P. Applying cognitive design principles to formatting HRQOL instruments. Qual Life Res. 2000;9:13-27 // Pesudovs K, Garamendi E, Keeves JP, Elliott DB. The Activities of Daily Vision Scale for cataract surgery outcomes: re-evaluating validity with Rasch analysis. Invest Ophthalmol Vis Sci 2003;44: 2892-9 // Pesudovs K, Garamendi E, Elliott DB. The Quality of Life Impact of Refractive Correction (QIRC) Questionnaire: develop¬ment and validation. Optom Vis Sci. 2004;81:769-777 // Pesudovs K, Burr JM, Harley C, Elliott DB. The development, assessment, and selection of questionnaires. Optom Vis Sci. 2007;84:663-74 // Pesudovs K, Ratcliffe J, Lamoureux EL, Lundström M, Massof RW, Rubin GS. Measuring the patient's perspective. Optom Vis Sci. 2013;90:717-9 // Revicki DA; Regulatory Issues and Patient-Reported Outcomes Task Force for the International Society for Quality of Life Research. FDA draft guidance and health-outcomes research. Lancet. 2007;369:540-2 // Schein OD. The measurement of patient-reported outcomes of refractive surgery: the refractive status and vision profile. Trans Am Ophthalmol Soc. 2000;98:439-469 // Sukhawarn R, Wiratchai N, Tatsanavivat P, Pitiyanuwat S, Kanato M, Srivannaboon S, Guyatt GH. Development of a refractive error quality of life scale for Thai adults (the REQ-Thai). J Med Assoc Thai. 2011;94:978-84 // Vandenbroeck S, De Geest S, Zeyen T, Stalmans I, Dobbels F. Patient-reported outcomes (PRO's) in glaucoma: a systematic review. Eye (Lond). 2011;25:555-77 // Vitale S, Schein OD, Meinert CL, Steinberg EP. The refractive status and vision profile: a questionnaire to measure vision-related quality of life in persons with refractive error. Ophthalmology. 2000;107:1529-1539